CLINICAL TRIAL: NCT04109066
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled Phase 3 Study of Nivolumab Versus Placebo in Combination With Neoadjuvant Chemotherapy and Adjuvant Endocrine Therapy in Patients With High-risk, Estrogen Receptor-Positive (ER+), Human Epidermal Growth Factor Receptor 2-Negative (HER2-) Primary Breast Cancer
Brief Title: Study of Nivolumab Versus Placebo in Combination With Neoadjuvant Chemotherapy and Adjuvant Endocrine Therapy in Participants With High-risk, Estrogen Receptor-Positive (ER+), Human Epidermal Growth Factor Receptor 2-Negative (HER2-) Primary Breast Cancer
Acronym: CheckMate 7FL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA209-7FL
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Nivolumab; Breast Cancer; Cancer; Estrogen Receptor-Positive (ER+); Human Epidermal Growth Factor 2 Negative (HER2-); Neoadjuvant; Adjuvant; Primary Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Nivolumab; Paclitaxel; Anthracyclines; Cyclophosphamide; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab combined with neoadjuvant CT and adjuvant ET (Experimental): Nivolumab with paclitaxel followed by nivolumab with anthracycline + cyclophosphamide as neoadjuvant (pre-surgery) treatment, then nivolumab with adjuvant (post-surgery) endocrine therapy of investigator's choice
  Interventions: Biological: nivolumab; Drug: paclitaxel (PTX); Drug: anthracycline; Drug: cyclophosphamide; Drug: Endocrine Therapy; Procedure: Surgery
- Arm B: Placebo combined with neoadjuvant CT and then adjuvant ET (Placebo Comparator): Nivolumab placebo with paclitaxel followed by nivolumab placebo with anthracycline + cyclophosphamide as neoadjuvant (pre-surgery) treatment, then adjuvant (post-surgery) endocrine therapy of investigator's choice
  Interventions: Drug: paclitaxel (PTX); Other: nivolumab placebo; Drug: anthracycline; Drug: cyclophosphamide; Drug: Endocrine Therapy; Procedure: Surgery

INTERVENTIONS:
Biological: nivolumab — Specified Dose on Specified days
  Arms: Arm A: Nivolumab combined with neoadjuvant CT and adjuvant ET
Drug: paclitaxel (PTX) — Specified dose on Specified days
Other: nivolumab placebo — Specified dose on Specified days
  Arms: Arm B: Placebo combined with neoadjuvant CT and then adjuvant ET
Drug: anthracycline — Specified dose on Specified days
Drug: cyclophosphamide — Specified dose on Specified days
Drug: Endocrine Therapy — Variable endocrine therapy of investigators choice
Procedure: Surgery — Surgery for breast cancer

SUMMARY:
A randomized multi-arm study evaluating the efficacy and safety of nivolumab versus placebo in combination with neoadjuvant (pre-surgery) chemotherapy and adjuvant (post-surgery) endocrine therapy in participants with high-risk, estrogen receptor-positive, human epidermal growth factor receptor 2-negative (ER+, HER2-) early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Localized invasive breast ductal carcinoma, confirmed by the local pathologist, that includes the following combined primary tumor and clinical node (cN) categories: T1c (tumor size = 2 cm)-T2 (tumor size > 2 cm), cN1-N2 OR T3-T4, cN0-cN2. Note: Axillary lymph node status must be assessed by fine needle biopsy or core biopsy.
* Estrogen receptor-positive (ER+) breast cancer (BC) and with or without progesterone receptor (PgR) expression (determined on the most recently analyzed tissue sample, tested locally, and confirmed by the central laboratory), as defined in the relevant American Society of Clinical Oncology (ASCO)- College of American Pathologists (CAP) Guidelines.
* Human epidermal growth factor receptor 2 (HER2-) BC tested in the local laboratory, defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0, 1+, or 2+.
* Tumor Grade 3 of ductal histology, Or Tumor Grade 2 of ductal histology having an ER expression level percentage between 1-10%
* Must agree to provide primary breast tumor tissue at baseline and at surgery
* Must be deemed eligible for surgery
* Males and females must agree to follow specific methods of contraception, if applicable, while participating in the trial
* Must have an Eastern Cooperative Oncology Group (ECOG) scale performance status of 0 or 1

Exclusion Criteria:

* Breastfeeding, pregnant, or expecting to conceive or father children within the projected duration of the study, starting with the screening through 12 months for participants who receive cyclophosphamide, or 6 months for participants who do not receive cyclophosphamide, after the last dose of study treatment
* Prior treatment with chemotherapy, endocrine therapy (ET), targeted therapy, and/or radiation therapy for the currently diagnosed breast cancer prior to enrollment
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Significant cardiovascular disease such as left ventricular ejection fraction (LVEF) < 50% at baseline as assessed by echocardiography (ECHO) or multigated acquisition (MUGA) scan performed at screening, or Class III or IV myocardial disease as described by the New York Heart Association
* History of ipsilateral invasive BC, regardless of treatment, ipsilateral ductal carcinoma in situ treated with radiation, or contralateral invasive BC, at any time
* Definitive clinical or radiologic evidence of metastatic disease
* Multicentric BC (the presence of > 1 tumor in different quadrants of the breast)
* Bilateral invasive BC

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (240):
- United States (30):
  - Local Institution - 0136, Mobile, Alabama
  - Local Institution - 0052, Greenbrae, California
  - Local Institution - 0051, Whittier, California
  - Local Institution - 0182, Stamford, Connecticut
  - Local Institution - 0150, Jacksonville, Florida
  - Local Institution - 0097, Miami, Florida
  - Local Institution - 0149, Pensacola, Florida
  - Local Institution - 0120, Tallahassee, Florida
  - Local Institution - 0054, Athens, Georgia
  - Local Institution - 0107, Atlanta, Georgia
  - Local Institution - 0056, Columbus, Georgia
  - Local Institution - 0221, Chicago, Illinois
  - Local Institution - 0227, Fort Wayne, Indiana
  - Local Institution - 0222, Topsham, Maine
  - Local Institution - 0146, Bethesda, Maryland
  - HCA Midwest Division, Kansas City, Missouri
  - Local Institution - 0109, Florham Park, New Jersey
  - Local Institution - 0050, Hackensack, New Jersey
  - Local Institution - 0180, New Brunswick, New Jersey
  - Local Institution - 0181, Albuquerque, New Mexico
  - Local Institution - 0041, The Bronx, New York
  - Local Institution - 0283, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Local Institution - 0053, Cleveland, Ohio
  - Local Institution - 0218, Nashville, Tennessee
  - Local Institution - 0121, Fort Worth, Texas
  - Local Institution - 0224, Fairfax, Virginia
  - Local Institution - 0122, Fredericksburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Local Institution - 0274, Seattle, Washington
- Argentina (12):
  - Local Institution - 0012, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Local Institution - 0015, La Plata, Buenos Aires
  - Local Institution - 0020, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0294, Córdoba, Córdoba Province
  - Local Institution - 0303, Río Cuarto, Córdoba Province
  - Local Institution - 0013, Buenos Aires, Distrito Federal
  - Local Institution - 0011, Caba, Distrito Federal
  - Local Institution - 0008, Capital Federal, Distrito Federal
  - Local Institution - 0014, Rosario Santa Fe, Santa Fe Province
  - Local Institution - 0021, Córdoba
  - Local Institution, La Rioja
  - Local Institution, Viedma
- Australia (8):
  - Local Institution - 0071, North Sydney, New South Wales
  - Local Institution - 0069, Port Macquarie, New South Wales
  - Local Institution - 0072, Herston, Queensland
  - Local Institution - 0067, Elizabeth Vale, South Australia
  - Local Institution - 0066, Clayton, Victoria
  - Local Institution - 0142, Clayton, Victoria
  - Local Institution - 0070, Melbourne, Victoria
  - Local Institution - 0068, North Ballarat, Victoria
- Austria (5):
  - Local Institution - 0045, Graz
  - Local Institution - 0042, Innsbruck
  - Local Institution - 0048, Salzburg
  - Local Institution - 0046, Vienna
  - Local Institution - 0047, Vienna
- Belgium (5):
  - Local Institution - 0187, Brussels
  - Local Institution - 0030, Charleroi
  - Local Institution - 0037, Edegem
  - Local Institution - 0032, Ghent
  - Local Institution - 0031, Liège
- Brazil (15):
  - Local Institution - 0130, Fortaleza, Ceará
  - Local Institution - 0225, Brasília, Federal District
  - Local Institution - 0287, Goiânia, Goiás
  - Local Institution - 0133, Belo Horizonte, Minas Gerais
  - Local Institution - 0132, Ijuí, Rio Grande do Sul
  - Local Institution - 0288, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0131, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0135, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0273, Santa Cruz do Sul, Rio Grande do Sul
  - Local Institution - 0134, Barretos, São Paulo
  - Local Institution - 0128, Santo André, São Paulo
  - Local Institution - 0272, São Paulo, São Paulo
  - Local Institution - 0129, Rio de Janeiro
  - Local Institution - 0144, São Paulo
  - Local Institution - 0104, São Paulo
- Canada (3):
  - Local Institution - 0095, Montreal, Quebec
  - Local Institution - 0194, Montreal, Quebec
  - Local Institution - 0058, Sherbrooke, Quebec
- Chile (6):
  - Local Institution - 0197, La Serena, Coquimbo Region
  - Local Institution - 0018, Viña del Mar, Región de Valparaíso
  - Local Institution - 0016, Santiago, Santiago Metropolitan
  - Local Institution - 0318, Santiago, Santiago Metropolitan
  - Local Institution - 0019, Santiago Region Metropolitana, Santiago Metropolitan
  - Local Institution - 0326, Antofagasta
- China (28):
  - Local Institution - 0235, Bengbu, Anhui
  - Local Institution - 0239, Hefei, Anhui
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution - 0319, Chongqing, Chongqing Municipality
  - Local Institution - 0232, Chongqing, Chongqing Municipality
  - Local Institution - 0267, Guangzhou, Guangdong
  - Local Institution - 0241, Guangzhou, Guangdong
  - Local Institution, Guangzhou, Guangdong
  - Local Institution - 0312, Zunyi, Guizhou
  - Local Institution - 0240, Shjiazhuang, Hebei
  - Local Institution - 0250, Wuhan, Hebei
  - Local Institution - 0248, Harbin, Heilongjiang
  - Local Institution, Zhengzhou, Henan
  - Local Institution - 0255, Changchun, Jilin
  - Local Institution - 0247, Changchun, Jilin
  - Local Institution - 0252, Shenyang, Liaoning
  - Local Institution - 0263, Xi'an, Shan3xi
  - Local Institution - 0245, Jinan, Shandong
  - Local Institution - 0256, Qingdao, Shandong
  - Local Institution - 0214, Yantai, Shandong
  - Local Institution - 0127, Shanghai, Shanghai Municipality
  - Local Institution - 0244, Chengdu, Sichuan
  - Local Institution - 0254, Tianjin, Tianjin Municipality
  - Local Institution - 0311, Ürümqi, Xinjiang
  - Local Institution - 0238, Hangzhou, Zhejiang
  - Local Institution - 0231, Hangzhou, Zhejiang
  - Local Institution - 0237, Hangzhou, Zhejiang
  - Local Institution - 0215, Beijing
- Colombia (8):
  - Local Institution - 0261, Barranquilla, Atlántico
  - Local Institution - 0094, Bogotá, Bogota D.C.
  - Local Institution - 0203, Colombia, Bogota D.C.
  - Local Institution - 0113, Montería, Departamento de Córdoba
  - Local Institution - 0098, Piedecuesta, Santander Department
  - Local Institution - 0093, Cali
  - Local Institution - 0271, Pereira
  - Local Institution - 0202, Rionegro
- Czechia (4):
  - Local Institution - 0100, Hradec Králové
  - Local Institution - 0103, Nový Jičín
  - Local Institution - 0101, Olomouc
  - Local Institution - 0099, Prague
- Denmark (4):
  - Local Institution - 0167, Aarhus N, Central Jutland
  - Local Institution - 0165, Herlev
  - Local Institution - 0164, København Ø
  - Local Institution - 0166, Næstved
- Finland (2):
  - Local Institution - 0001, Helsinki
  - Local Institution - 0160, Tampere
- France (12):
  - Local Institution - 0216, Le Mans, Sarthe
  - Local Institution - 0004, Besançon
  - Local Institution - 0024, Brest
  - Local Institution - 0162, Clermont-Ferrand
  - Local Institution - 0153, Lyon
  - Local Institution - 0152, Montpellier
  - Local Institution - 0161, Paris
  - Local Institution - 0195, Plérin
  - Local Institution - 0002, Saint-Herblain
  - Local Institution - 0258, Strasbourg
  - Local Institution - 0228, Toulon
  - Local Institution - 0003, Villejuif
- Germany (15):
  - Local Institution - 0084, München, Bavaria
  - Local Institution - 0079, Saarbrücken, Saarland
  - Local Institution - 0083, Berlin
  - Local Institution - 0080, Cologne
  - Local Institution - 0112, Dresden
  - Local Institution - 0081, Essen
  - Local Institution - 0158, Frankfurt
  - Local Institution - 0223, Hamburg
  - Local Institution - 0087, Heidelberg
  - Local Institution - 0089, Homburg
  - Local Institution - 0196, Leipzig
  - Local Institution - 0111, Mönchengladbach
  - Local Institution - 0156, Rostock
  - Local Institution - 0157, Velbert
  - Local Institution - 0105, Würzburg
- Local Institution - 0115, Hong Kong, Hong Kong
- Ireland (3):
  - Local Institution - 0034, Dublin, Dublin
  - Local Institution - 0035, Beaumont
  - Local Institution - 0036, Cork
- Italy (8):
  - Local Institution - 0191, Catanzaro
  - Local Institution - 0207, Milan
  - Azienda Ospedaliero Universitaria Federico II di Napoli, Napoli
  - Local Institution - 0124, Napoli
  - Local Institution - 0155, Padua
  - Fondazione Irccs - Policlinico San Matteo, Pavia
  - Local Institution - 0190, Roma
  - Local Institution - 0125, Rozzano (MI)
- Mexico (10):
  - Local Institution - 0262, Tijuana, Estado de Baja California
  - Local Institution - 0330, Zapopan, Jalisco
  - Local Institution - 0168, Mexico City, Mexico City
  - Local Institution - 0154, Mexico City, Mexico City
  - Local Institution - 0137, Monterrey, Nuevo León
  - Local Institution - 0212, Mérida, Yucatán
  - Local Institution - 0280, Campeche
  - Local Institution - 0091, Chihuahua City
  - Local Institution - 0145, Colima
  - Local Institution - 0141, Oaxaca City
- Netherlands (4):
  - Local Institution - 0033, Amsterdam
  - Local Institution - 0177, Breda
  - Local Institution - 0199, Deventer
  - Local Institution - 0147, Utrecht
- Poland (7):
  - Local Institution - 0334, Gliwice, Silesian Voivodeship
  - Local Institution - 0335, Bydgoszcz
  - Local Institution - 0061, Koszalin
  - Local Institution - 0059, Krakow
  - Local Institution - 0063, Lodz
  - Local Institution - 0062, Opole
  - Local Institution - 0060, Warsaw
- Portugal (3):
  - Local Institution - 0210, Lisbon
  - Local Institution - 0211, Lisbon
  - Local Institution - 0209, Porto
- Local Institution - 0110, Ponce, Puerto Rico
- Romania (6):
  - Local Institution - 0029, Bucharest
  - Local Institution - 0025, Bucharest
  - Local Institution - 0270, Bucharest
  - Local Institution - 0028, Craiova
  - Local Institution - 0027, Floreşti
  - Local Institution - 0026, Suceava
- Russia (8):
  - Local Institution, Krasnodar
  - Local Institution - 0119, Moscow
  - Local Institution, Moscow
  - Local Institution - 0285, Moskva
  - Local Institution, Ryazan
  - Local Institution - 0306, Saint Petersburg
  - Local Institution - 0284, Saint Petersburg
  - Local Institution, Sochi
- Singapore (3):
  - Local Institution - 0078, Singapore
  - Local Institution - 0076, Singapore
  - Local Institution - 0077, Singapore
- South Korea (5):
  - Local Institution - 0325, Seongnam
  - Local Institution - 0295, Seoul
  - Local Institution - 0320, Seoul
  - Local Institution - 0290, Seoul
  - Local Institution - 0291, Seoul
- Spain (10):
  - Local Institution - 0205, Elche, Alicante
  - Local Institution - 0171, Barcelona
  - Local Institution - 0172, Barcelona
  - Local Institution - 0173, Madrid
  - Local Institution - 0176, Madrid
  - Local Institution - 0169, Málaga
  - Local Institution - 0204, Pamplona
  - Local Institution - 0174, Santiago de Compostela
  - Local Institution - 0170, Seville
  - Local Institution - 0175, Valencia
- Switzerland (3):
  - Local Institution - 0184, Basel
  - Local Institution - 0186, Lausanne
  - Local Institution - 0185, Thun
- Taiwan (5):
  - Local Institution - 0301, Kaohsiung City
  - Local Institution - 0298, Tainan
  - Local Institution - 0300, Tainan
  - Local Institution - 0305, Taipei
  - Local Institution - 0297, Taipei
- Turkey (Türkiye) (4):
  - Local Institution - 0073, Adana
  - Local Institution - 0257, Ankara
  - Local Institution - 0075, Antalya
  - Local Institution - 0074, Istanbul
- United Kingdom (2):
  - Local Institution - 0006, Withington, Manchester
  - Local Institution - 0005, London

REFERENCES:
- [Derived] Loi S, Salgado R, Curigliano G, Romero Diaz RI, Delaloge S, Rojas Garcia CI, Kok M, Saura C, Harbeck N, Mittendorf EA, Yardley DA, Suarez Zaizar A, Caminos FR, Ungureanu A, Reinoso-Toledo JG, Guarneri V, Egle D, Ades F, Pacius M, Chhibber A, Chandra R, Nathani R, Spires T, Wu JQ, Pusztai L, McArthur H. Neoadjuvant nivolumab and chemotherapy in early estrogen receptor-positive breast cancer: a randomized phase 3 trial. Nat Med. 2025 Feb;31(2):433-441. doi: 10.1038/s41591-024-03414-8. Epub 2025 Jan 21. PMID 39838118
- [Derived] Schlam I, Corti C, Sammons S, Mittendorf EA, Tolaney SM. Checkpoint inhibition for early-stage hormone receptor-positive breast cancer. Expert Opin Biol Ther. 2024 Jun;24(6):511-520. doi: 10.1080/14712598.2024.2370395. Epub 2024 Jun 24. PMID 38913933
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 Participants planned for Arm B treatment received Arm A treatment.
Groups:
- Arm A: Neoadjuvant (Pre-surgery) Phase 8 cycles maximum:
  Paclitaxel (PTX) Cycles 1-4 (1 cycle = Q3W): Nivolumab 360 mg Q3W + PTX QW
  Followed by:
  Anthracycline-Cyclophosphamide (AC) Cycles 1-4 (1 cycle = Q2W or Q3W):
  Nivolumab 360 mg Q3W + AC Q3W or Nivolumab 240 mg Q2W + AC Q2W
  Surgery and Adjuvant (Post-surgery) Phase 7 cycles maximum:
  Adjuvant Cycles 1-7 (1 cycle = Q4W):
  Nivolumab 480 mg Q4W + Endocrine Therapy (ET)
- Arm B: Neoadjuvant (Pre-surgery) Phase 8 cycles maximum:
  Paclitaxel (PTX) Cycles 1-4 (1 cycle = Q3W): Nivolumab Placebo Q3W + PTX QW
  Followed by:
  Anthracycline-Cyclophosphamide (AC) Cycles 1-4 (1 cycle = Q2W or Q3W):
  Nivolumab Placebo Q3W + AC Q3W or Nivolumab Placebo Q2W + AC Q2W
  Surgery and Adjuvant (Post-surgery) Phase 7 cycles maximum:
  Adjuvant Cycles 1-7 (1 cycle = Q4W):
  Endocrine Therapy (ET)
Period: Pre-treatment
Arm/Group | Arm A | Arm B
Started (Started = Randomized) | 263 | 258
Completed (Completed = Treated) | 260 | 257
Not Completed | 3 | 1
Not completed — Participant withdrew consent | 2 | 0
Not completed — Participant no longer meets study criteria | 1 | 1
Period: Treatment
Arm/Group | Arm A | Arm B
Started (Started = Treated) | 260 | 257
Received Arm A Treatment | 0 | 2 (Planned for Arm B treatment but received Arm A treatment.)
Completed | 167 | 174
Not Completed | 93 | 83
Not completed — Lack of Efficacy | 2 | 4
Not completed — Adverse Event | 23 | 7
Not completed — Participant request to discontinue Study treatment | 15 | 14
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Death | 3 | 0
Not completed — Participant no longer meets study criteria | 2 | 2
Not completed — Administrative reasons by sponsor | 2 | 3
Not completed — Other reasons | 17 | 23
Not completed — Disease Progression | 4 | 7
Not completed — Study drug toxicity | 12 | 5
Not completed — Adverse Event unrelated to Study drug | 1 | 0
Not completed — Disease Recurrence | 0 | 2
Not completed — Not reported | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 263 | 258 | 521
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12.0) | 50.9 (11.8) | 50.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262 | 257 | 519
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 80 | 154
  Not Hispanic or Latino | 102 | 121 | 223
  Unknown or Not Reported | 87 | 57 | 144
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 17 | 35
  Asian | 24 | 18 | 42
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 6 | 8 | 14
  White | 202 | 193 | 395
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 19 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: pCR rate is defined as the percentage of participants who achieved pCR. pCR is defined as no invasive residual disease in breast and lymph nodes performed by a local pathologist. Criteria for evaluation of pCR includes the following: pCR in breast, axillary lymph nodes and non-axillary sentinel node; no histologic evidence of invasive tumor cells; and pCR in the breast.
Time Frame: Up to approximately 37 months
Population: All randomized participants with sufficient follow-up for pCR assessment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 257 | 253
Percentage of participants | 24.5 [19.4 to 30.2] | 13.8 [9.8 to 18.7]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Arm A over Arm B; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.29 to 3.27] — Stratified by PD-L1 by SP142 (< 1% vs. >= 1%), AC Dose-Frequency Chemotherapy Regimen (Q2W vs. Q3W) per IRT. Strata adjusted odds ratio (Arm A over Arm B) using Mantel-Haenszel method
Statistical Analysis 2: Comparison: Arm A vs Arm B; Test type: Other; Adjusted Difference of pCR Rates = 10.5, 95% CI 2-sided [4.0 to 16.9] — Strata adjusted difference in pCR (Arm A-B) based on Cochran-Mantel-Haenszel (CMH) method of weighting. Stratified by PD-L1 by SP142 (< 1% vs. >= 1%), AC Dose-Frequency Chemotherapy Regimen (Q2W vs. Q3W) per IRT

2. Secondary Outcome: Pathological Complete Response (pCR) Rate (PD-L1 >=1%)
Description: as for outcome 1
Time Frame: Up to approximately 37 months
Population: All randomized participants in PD-L1 expression on immune cells >=1% subgroup with sufficient follow-up for pCR assessment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 88 | 84
Percentage of participants | 44.3 [33.7 to 55.3] | 20.2 [12.3 to 30.4]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Arm A over Arm B; Test type: Superiority; Odds Ratio (OR) = 3.11, 95% CI 2-sided [1.58 to 6.11] — Stratified by AC Dose-Frequency. Chemotherapy Regimen (Q2W vs. Q3W) per IRT. Strata adjusted odds ratio (Arm A over Arm B) using Mantel-Haenszel method
Statistical Analysis 2: Comparison: Arm A vs Arm B; Test type: Other; Adjusted Difference of pCR Rates = 24.1, 95% CI 2-sided [10.7 to 37.5] — Strata adjusted difference in pCR (Arm A-B) based on Cochran-Mantel-Haenszel (CMH) method of weighting. Stratified by AC Dose-Frequency Chemotherapy Regimen (Q2W vs. Q3W) per IRT

3. Secondary Outcome: Number of Participants With Residual Cancer Burden (RCB)
Description: RCB is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. RCB is categorized into the following 4 classes: RCB-0: no residual disease; RCB-1: minimal residual disease; RCB-II: moderate residual disease; RCB-III: and extensive residual disease.
Time Frame: Up to approximately 37 months
Population: All randomized participants with sufficient follow-up for RCB assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 257 | 253
Participants
  RCB-0 | 62 | 34
  RCB-I | 17 | 20
  RCB-II | 90 | 106
  RCB-III | 57 | 73
  Not Reported | 31 | 20

4. Secondary Outcome: Number of Participants With Residual Cancer Burden (RCB) PD-L1 >=1%
Description: as for outcome 3
Time Frame: Up to approximately 37 months
Population: All randomized participants in PD-L1 expression on immune cells >=1% subgroup with sufficient follow-up for RCB assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 88 | 84
Participants
  RCB-0 | 38 | 16
  RCB-I | 10 | 6
  RCB-II | 25 | 36
  RCB-III | 9 | 20
  Not Reported | 6 | 6

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with any grade adverse events (AEs). An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relation with this treatment. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: From first dose to 30 days post last dose of neoadjuvant or adjuvant study therapy (Up to approximately 19 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 262 | 255
Participants
  Adverse Events (AEs) | 259 | 252
  Drug-Related AEs | 254 | 236
  AEs leading to discontinuation | 41 | 14

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with any grade serious adverse events (SAE). SAE is defined as any untoward medical occurrence that, at any dose: Results in death; is life threatening; requires inpatient hospitalization; results in persistent or significant disability; is a congenital anomaly/birth defect. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: From first dose to 30 days post last dose of neoadjuvant or adjuvant study therapy (Up to approximately 19 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 262 | 255
Participants | 80 | 45

7. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died due to any cause.
Time Frame: Up to approximately 41 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 262 | 255
Participants | 15 | 8

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 41 months). SAEs and Other AEs were assessed from first dose up to 100 days post last dose (Up to approximately 21 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants based on the treatment received. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
  The 2 participants planned for Arm B treatment but received Arm A treatment are accounted for in the Arm A groups.
Groups:
- Arm A: Nivo + Chemo (PTX QW + AC Q3W) / Nivo + ET: Neoadjuvant (Pre-surgery) Phase 8 cycles maximum:
  Paclitaxel (PTX) Cycles 1-4 (1 cycle = Q3W): Nivolumab 360 mg Q3W + PTX QW
  Followed by:
  Anthracycline-Cyclophosphamide (AC) Cycles 1-4 (1 cycle = Q3W):
  Nivolumab 360 mg Q3W + AC Q3W
  Surgery and Adjuvant (Post-surgery) Phase 7 cycles maximum:
  Adjuvant Cycles 1-7 (1 cycle = Q4W):
  Nivolumab 480 mg Q4W + Endocrine Therapy (ET)
- Arm A: Nivo + Chemo (PTX QW + AC Q2W) / Nivo + ET: Neoadjuvant (Pre-surgery) Phase 8 cycles maximum:
  Paclitaxel (PTX) Cycles 1-4 (1 cycle = Q3W): Nivolumab 360 mg Q3W + PTX QW
  Followed by:
  Anthracycline-Cyclophosphamide (AC) Cycles 1-4 (1 cycle = Q2W):
  Nivolumab 240 mg Q2W + AC Q2W
  Surgery and Adjuvant (Post-surgery) Phase 7 cycles maximum:
  Adjuvant Cycles 1-7 (1 cycle = Q4W):
  Nivolumab 480 mg Q4W + Endocrine Therapy (ET)
- Arm B: Nivo Placebo + Chemo (PTX QW + AC Q3W) / ET: Neoadjuvant (Pre-surgery) Phase 8 cycles maximum:
  Paclitaxel (PTX) Cycles 1-4 (1 cycle = Q3W): Nivolumab Placebo Q3W + PTX QW
  Followed by:
  Anthracycline-Cyclophosphamide (AC) Cycles 1-4 (1 cycle = Q3W):
  Nivolumab Placebo Q3W + AC Q3W
  Surgery and Adjuvant (Post-surgery) Phase 7 cycles maximum:
  Adjuvant Cycles 1-7 (1 cycle = Q4W):
  Endocrine Therapy (ET)
- Arm B: Nivo Placebo + Chemo (PTX QW + AC Q2W) / ET: Neoadjuvant (Pre-surgery) Phase 8 cycles maximum:
  Paclitaxel (PTX) Cycles 1-4 (1 cycle = Q3W): Nivolumab Placebo Q3W + PTX QW
  Followed by:
  Anthracycline-Cyclophosphamide (AC) Cycles 1-4 (1 cycle = Q2W):
  Nivolumab Placebo Q2W + AC Q2W
  Surgery and Adjuvant (Post-surgery) Phase 7 cycles maximum:
  Adjuvant Cycles 1-7 (1 cycle = Q4W):
  Endocrine Therapy (ET)
Arm/Group | Arm A: Nivo + Chemo (PTX QW + AC Q3W) / Nivo + ET | Arm A: Nivo + Chemo (PTX QW + AC Q2W) / Nivo + ET | Arm B: Nivo Placebo + Chemo (PTX QW + AC Q3W) / ET | Arm B: Nivo Placebo + Chemo (PTX QW + AC Q2W) / ET
All-Cause Mortality (participants affected / at risk) | 8/129 | 7/136 | 4/124 | 4/132
Serious Adverse Events (participants affected / at risk) | 38/127 | 51/135 | 20/123 | 26/132
Other Adverse Events (participants affected / at risk) | 126/127 | 132/135 | 120/123 | 130/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivo + Chemo (PTX QW + AC Q3W) / Nivo + ET (N=127) | Arm A: Nivo + Chemo (PTX QW + AC Q2W) / Nivo + ET (N=135) | Arm B: Nivo Placebo + Chemo (PTX QW + AC Q3W) / ET (N=123) | Arm B: Nivo Placebo + Chemo (PTX QW + AC Q2W) / ET (N=132)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 9 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac perfusion defect (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 1 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0
Immune-mediated adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Thyroiditis subacute (Endocrine disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Death (General disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 4 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 2 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 5 | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 3 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 1 | 1
Neutropenic infection (Infections and infestations) | 0 | 1 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 1 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 2 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
SARS-CoV-2 sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1
Systemic infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Vascular access site infection (Infections and infestations) | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Surgical procedure repeated (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Inflammatory marker increased (Investigations) | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Breast inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivo + Chemo (PTX QW + AC Q3W) / Nivo + ET (N=127) | Arm A: Nivo + Chemo (PTX QW + AC Q2W) / Nivo + ET (N=135) | Arm B: Nivo Placebo + Chemo (PTX QW + AC Q3W) / ET (N=123) | Arm B: Nivo Placebo + Chemo (PTX QW + AC Q2W) / ET (N=132)
Anaemia (Blood and lymphatic system disorders) | 47 | 65 | 32 | 62
Leukopenia (Blood and lymphatic system disorders) | 8 | 8 | 12 | 11
Lymphopenia (Blood and lymphatic system disorders) | 15 | 9 | 8 | 12
Neutropenia (Blood and lymphatic system disorders) | 24 | 26 | 27 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 7 | 1 | 3
Palpitations (Cardiac disorders) | 2 | 6 | 1 | 7
Tachycardia (Cardiac disorders) | 3 | 8 | 0 | 4
Adrenal insufficiency (Endocrine disorders) | 5 | 10 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 7 | 13 | 2 | 5
Hypothyroidism (Endocrine disorders) | 19 | 30 | 8 | 5
Dry eye (Eye disorders) | 4 | 10 | 4 | 11
Lacrimation increased (Eye disorders) | 4 | 7 | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 15 | 9 | 12
Abdominal pain upper (Gastrointestinal disorders) | 7 | 12 | 4 | 9
Constipation (Gastrointestinal disorders) | 23 | 36 | 19 | 30
Diarrhoea (Gastrointestinal disorders) | 30 | 48 | 26 | 40
Dry mouth (Gastrointestinal disorders) | 5 | 9 | 4 | 7
Dyspepsia (Gastrointestinal disorders) | 9 | 10 | 5 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 9 | 2 | 14
Nausea (Gastrointestinal disorders) | 61 | 77 | 55 | 59
Stomatitis (Gastrointestinal disorders) | 4 | 14 | 4 | 12
Vomiting (Gastrointestinal disorders) | 26 | 27 | 25 | 13
Asthenia (General disorders) | 27 | 25 | 30 | 27
Chills (General disorders) | 1 | 8 | 1 | 2
Fatigue (General disorders) | 34 | 67 | 24 | 52
Illness (General disorders) | 7 | 0 | 2 | 1
Mucosal inflammation (General disorders) | 7 | 16 | 6 | 19
Oedema peripheral (General disorders) | 5 | 12 | 6 | 13
Pain (General disorders) | 5 | 11 | 2 | 3
Pyrexia (General disorders) | 11 | 21 | 7 | 10
Hypersensitivity (Immune system disorders) | 8 | 3 | 5 | 8
COVID-19 (Infections and infestations) | 21 | 29 | 18 | 29
Folliculitis (Infections and infestations) | 6 | 9 | 1 | 5
Nasopharyngitis (Infections and infestations) | 4 | 6 | 1 | 7
Upper respiratory tract infection (Infections and infestations) | 1 | 7 | 8 | 5
Urinary tract infection (Infections and infestations) | 12 | 8 | 9 | 11
Infusion related reaction (Injury, poisoning and procedural complications) | 12 | 25 | 10 | 12
Procedural pain (Injury, poisoning and procedural complications) | 3 | 9 | 5 | 5
Radiation skin injury (Injury, poisoning and procedural complications) | 15 | 22 | 13 | 20
Alanine aminotransferase increased (Investigations) | 27 | 31 | 23 | 20
Aspartate aminotransferase increased (Investigations) | 32 | 30 | 23 | 19
Blood alkaline phosphatase increased (Investigations) | 10 | 9 | 4 | 5
Blood calcium increased (Investigations) | 0 | 7 | 0 | 3
Blood glucose increased (Investigations) | 0 | 7 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 6 | 6 | 5 | 9
Blood sodium decreased (Investigations) | 0 | 8 | 0 | 5
Blood thyroid stimulating hormone decreased (Investigations) | 4 | 11 | 0 | 3
Blood thyroid stimulating hormone increased (Investigations) | 5 | 15 | 3 | 4
Lymphocyte count decreased (Investigations) | 4 | 9 | 2 | 3
Neutrophil count decreased (Investigations) | 20 | 16 | 11 | 11
Weight decreased (Investigations) | 7 | 10 | 3 | 3
White blood cell count decreased (Investigations) | 15 | 9 | 8 | 5
Decreased appetite (Metabolism and nutrition disorders) | 16 | 19 | 13 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 13 | 8 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 12 | 0 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 2 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 41 | 20 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 16 | 5 | 17
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 12 | 4 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 26 | 13 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 14 | 8 | 12
Dizziness (Nervous system disorders) | 9 | 10 | 7 | 8
Dysgeusia (Nervous system disorders) | 9 | 26 | 8 | 14
Headache (Nervous system disorders) | 24 | 43 | 24 | 33
Neuropathy peripheral (Nervous system disorders) | 26 | 38 | 19 | 32
Paraesthesia (Nervous system disorders) | 8 | 10 | 8 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 21 | 10 | 16
Taste disorder (Nervous system disorders) | 0 | 3 | 1 | 9
Anxiety (Psychiatric disorders) | 6 | 10 | 2 | 6
Depression (Psychiatric disorders) | 3 | 7 | 0 | 8
Insomnia (Psychiatric disorders) | 8 | 25 | 8 | 20
Breast pain (Reproductive system and breast disorders) | 4 | 13 | 6 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 29 | 9 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 9 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 8 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 4 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 83 | 64 | 80 | 69
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 7 | 3 | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 10 | 10 | 9
Onycholysis (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 22 | 5 | 18
Rash (Skin and subcutaneous tissue disorders) | 18 | 30 | 16 | 28
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 8
Flushing (Vascular disorders) | 0 | 7 | 3 | 7
Hot flush (Vascular disorders) | 9 | 33 | 12 | 30
Hypertension (Vascular disorders) | 11 | 9 | 5 | 7
Lymphoedema (Vascular disorders) | 2 | 5 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT04109066/Prot_SAP_000.pdf